CLINICAL TRIAL: NCT06628063
Title: Second and Third Trimestric Scan Versus Second Trimestric Scan Alone in Detection of Congenital Fetal Anomalies
Brief Title: Examination of Pregnant Women in Third Trimester by Ultrasound to Detect Any Congenital Anomalies
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Desouky, Resident, Sohag University
Other Study IDs: soh -Med-24-09-16MS
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Congenital Anomaly
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal third trimestric scam: cases in which second and third trimestric scan show no additional benefit over second trimestric scan alone
  Interventions: Other: ultrasound evaluation
- new finding in third trimestric scan: cases in which second and third trimestric scan show additional benefit over second trimestric scan alone
  Interventions: Other: ultrasound evaluation

INTERVENTIONS:
Other: ultrasound evaluation — Ultrasound scan of fetus in second and third trimestrers

SUMMARY:
this study aims to help the physicians to evaluate the practice of routine Third trimestric fetal scan whether it should be routinely performed to all cases including those with low risk singleton pregnancies.

DETAILED DESCRIPTION:
The third-trimester ultrasound scan ,traditionally performed at 32-34weeks, can assess fetal viability , presentation, anatomy , growth, amniotic fluid volume, placental location and fetoplacental Doppler.

There are multiple other indications that can trigger a third-trimester scan, including antepartum bleeding , reduced fetal movements, preterm rupture of the membranes and suspected abnormalities of fetal growth based on physical examination. In addition, ultrasound may be used to guide other procedures in the third trimester, such as external cephalic version. However, as yet, there is no convincing evidence that routine universal third-trimester ultrasound examination in a low-risk population improves either perinatal or maternal outcome especially in low socioeconomic countries with limited resources

ELIGIBILITY:
Inclusion Criteria:

* Singleton healthy pregnancy at second and third trimesters of pregnancy.
* Fetuses were considered normal based on second trimestric fetal scan in our feto-maternal unit

Exclusion Criteria:

* Exclusion criteria were patients with multiple gestations, maternal medical complications as Preeclampsia, DM ,Cardiac or renal diseases , or fetal abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant female at second trimester
Study Population: normal pregnancies attending outpatient clinic in Sohag university Hospital
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
newly discovered congenital anomaly at third trimester of pregnancy | from October 2024 to April 2025
  assessing Additional benefit of 3rd Trimester scan in low risk pregnancies attending sohag university regarding detection pf fetal congenital anomalies

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud desoky Desoky, Principal Investigator — sohag university , Department of obstetric and gynecology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Guidelines from international society of ultrasound about fetal scanning at third trimester — https://www.isuog.org/resource/isuog-practice-guidelines-performance-of-third-trimester-obstetric.html